CLINICAL TRIAL: NCT00014612
Title: After Mapping Of The Axilla: Radiotherapy Or Surgery
Brief Title: Comparison of Complete Axillary Lymph Node Dissection With Axillary Radiation Therapy in Treating Women With Invasive Breast Cancer
Acronym: AMAROS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: ALMANAC Trialists Group (Unknown); Borstkanker Onderzoeksgroup Nederland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-10981-22023
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

ARMS (2):
- axillary lymph node dissection (Active Comparator): complete axillary lymph node dissection
  Interventions: Procedure: axillary lymph node dissection; Procedure: lymphoscintigraphy; Procedure: therapeutic conventional surgery
- axillary radiotherapy (Experimental): axillary radiotherapy, daily for 5 days a week, for 5 weeks
  Interventions: Procedure: lymphoscintigraphy; Procedure: therapeutic conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Procedure: axillary lymph node dissection
  Arms: axillary lymph node dissection
Procedure: lymphoscintigraphy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy
  Arms: axillary radiotherapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells and may be a less invasive treatment and cause fewer side effects than complete axillary lymph node dissection. It is not yet known which treatment is more effective for invasive breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of complete axillary lymph node dissection with that of axillary radiation therapy in treating women who have invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the regional control of the axilla obtained by complete axillary lymph node dissection vs axillary radiotherapy in sentinel lymph node-positive women with operable invasive breast cancer.
* Determine whether local and regional axillary control can be obtained without axillary lymph node dissection in sentinel lymph node-negative women.
* Compare the axillary 5-year recurrence-free survival of these patients treated with these regimens.
* Compare the morbidity of patients treated with these regimens.
* Compare the quality of life of these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and type of breast surgery (conservation vs total mastectomy). Patients are randomized to 1 of 2 treatment arms.

Patients are given an injection of a tracer and undergo lymphoscintigraphy 2-3 hours later to identify the sentinel lymph node. Within 24 hours after lymphoscintigraphy, patients undergo wide local excision of the tumor or mastectomy after the sentinel node is removed. If no sentinel node is found or metastasis is found in a nonsentinel node, patients undergo complete axillary lymph node dissection (ALND) regardless of randomization. Sentinel node-negative patients receive no further treatment. Sentinel node-positive patients continue treatment according to randomization.

* Arm I: Within 8 weeks after surgery, patients undergo complete ALND.
* Arm II: Within 8 weeks after surgery, patients undergo axillary lymph node radiotherapy daily 5 days a week for 5 weeks.

Patients in arm I may receive postoperative axillary irradiation if 4 or more nodes are positive and more than 1 axillary level is involved.

Quality of life is assessed at baseline and then at 1, 2, 3, and 5 years.

Patients are followed annually for 5 years.

PROJECTED ACCRUAL: A total of 3,485 patients (1,394 sentinel node-positive and 2,091 sentinel node-negative) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or "triple diagnosis" (palpation, mammogram or ultrasound, and cytology) confirmed operable invasive breast cancer

  * T0-2, N0
  * Diagnosis by excisional tumorectomy allowed
  * Clinically occult invasive disease must be histologically confirmed
* Only 1 tumor in 1 breast

  * Tumor between 5 and 50 mm in largest diameter, within 1 quadrant by mammogram, ultrasound or MRI

    * Multifocal (i.e., within one quadrant and sharing the same histological characteristics) is allowed
    * Multicentric (i.e., in different quadrants) breast cancer is not allowed
* Clinically negative axillary lymph nodes
* No metastatic disease
* No previous treatment of the primary breast tumor by neoadjuvant hormonal or systemic treatment
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Any age

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Fit to undergo sentinel node biopsy, axillary clearance, breast surgery, and/or axillary radiotherapy
* No psychological, familial, sociological, or geographical condition that would preclude study compliance
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to axilla

Surgery:

* No prior surgery to axilla

Other:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4813 (Actual)
Dates: Start 2001-02; Primary Completion 2010-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Axillary recurrence rate | from randomization

SECONDARY OUTCOMES:
Shoulder function as assessed by arm function test questionnaire at baseline, 1, 3, and 5 years after surgery | from randomization
Quality of life as measured by Quality of Life Questionnaire Core 30 Items (QLQ-C30) and QLQ-BR25 at baseline, 1, 2, 3, and 5 years after surgery | from randomization
Axillary recurrence-free survival | from randomization
Disease-free survival | from randomization
Overall survival | from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Emiel JT Rutgers, Study Chair — The Netherlands Cancer Institute; Robert Mansel, Study Chair — Cardiff and Vale University Health Board - University Hospital of Wales, Cardiff; Cornelis Van De Velde, Study Chair — Leiden University Medical Centre, Leiden; Geertjan Van Tienhoven, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam, Amsterdam
Locations (29):
- France (2):
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Oscar Lambret, Lille
- Italy (2):
  - Universita Degli Studi di Florence - Policlinico di Careggi, Firenze (Florence)
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
- Netherlands (19):
  - Ziekenhuis Amstelland, Amstelveen
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Gelre Ziekenhuizen - Lokatie Lukas, Apeldoorn
  - Rijnstate Hospital, Arnhem
  - Reinier de Graaf Group - Delft, Delft
  - NIJ Smellinghe, Drachten
  - Catharina Ziekenhuis, Eindhoven
  - University Medical Center Groningen, Groningen
  - Kennemer Gasthuis - Locatie EG, Haarlem
  - Ropcke-Zweers Ziekenhuis, Hardenberg
  - Ziekenhuis St. Jansdal, Harderwijk
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Saint Laurentius Ziekenhuis, Roermond
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
  - HagaZiekenhuis - Locatie Rode Kruis, The Hague
  - Ziekenhuis Bronovo, The Hague
  - University Medical Center Utrecht, Utrecht
- Medical University of Gdansk, Gdansk, Poland
- Institute of Oncology - Ljubljana, Ljubljana, Slovenia
- Hopital Cantonal Universitaire de Geneve, Geneva, Switzerland
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Wythenshawe Hospital, Manchester, England
  - University Hospital of Wales, Cardiff, Wales

REFERENCES:
- [Result] Straver ME, Meijnen P, van Tienhoven G, van de Velde CJ, Mansel RE, Bogaerts J, Demonty G, Duez N, Cataliotti L, Klinkenbijl J, Westenberg HA, van der Mijle H, Hurkmans C, Rutgers EJ. Role of axillary clearance after a tumor-positive sentinel node in the administration of adjuvant therapy in early breast cancer. J Clin Oncol. 2010 Feb 10;28(5):731-7. doi: 10.1200/JCO.2008.21.7554. Epub 2009 Dec 28. PMID 20038733
- [Result] Straver ME, Meijnen P, van Tienhoven G, van de Velde CJ, Mansel RE, Bogaerts J, Duez N, Cataliotti L, Klinkenbijl JH, Westenberg HA, van der Mijle H, Snoj M, Hurkmans C, Rutgers EJ. Sentinel node identification rate and nodal involvement in the EORTC 10981-22023 AMAROS trial. Ann Surg Oncol. 2010 Jul;17(7):1854-61. doi: 10.1245/s10434-010-0945-z. Epub 2010 Mar 19. PMID 20300966
- [Result] Straver ME, Meijnen P, van Tienhoven G, et al.: Technical aspects of the sentinel node biopsy in the EORTC AMAROS sentinel node trial. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-1006, 2008.
- [Result] Meijnen P, Rutgers EJT, van de Velde CJH, et al.: EORTC 10981-22023 trial. AMAROS: after mapping of the axilla: radiotherapy or surgery? Trial update. [Abstract] Eur J Cancer 2 (Suppl 3): A-79, 79, 2004.
- [Result] Hurkmans CW, Borger JH, Rutgers EJ, van Tienhoven G; EORTC Breast Cancer Cooperative Group; Radiotherapy Cooperative Group. Quality assurance of axillary radiotherapy in the EORTC AMAROS trial 10981/22023: the dummy run. Radiother Oncol. 2003 Sep;68(3):233-40. doi: 10.1016/s0167-8140(03)00194-4. PMID 13129630
- [Derived] Donker M, Slaets L, van Tienhoven G, Rutgers EJ. [Axillary lymph node dissection versus axillary radiotherapy in patients with a positive sentinel node: the AMAROS trial]. Ned Tijdschr Geneeskd. 2015;159:A9302. Dutch. PMID 26488192
- [Derived] Donker M, van Tienhoven G, Straver ME, Meijnen P, van de Velde CJ, Mansel RE, Cataliotti L, Westenberg AH, Klinkenbijl JH, Orzalesi L, Bouma WH, van der Mijle HC, Nieuwenhuijzen GA, Veltkamp SC, Slaets L, Duez NJ, de Graaf PW, van Dalen T, Marinelli A, Rijna H, Snoj M, Bundred NJ, Merkus JW, Belkacemi Y, Petignat P, Schinagl DA, Coens C, Messina CG, Bogaerts J, Rutgers EJ. Radiotherapy or surgery of the axilla after a positive sentinel node in breast cancer (EORTC 10981-22023 AMAROS): a randomised, multicentre, open-label, phase 3 non-inferiority trial. Lancet Oncol. 2014 Nov;15(12):1303-10. doi: 10.1016/S1470-2045(14)70460-7. Epub 2014 Oct 15. PMID 25439688
- [Derived] Donker M, Straver ME, van Tienhoven G, van de Velde CJ, Mansel RE, Litiere S, Werutsky G, Duez NJ, Orzalesi L, Bouma WH, van der Mijle H, Nieuwenhuijzen GA, Veltkamp SC, Helen Westenberg A, Rutgers EJ. Comparison of the sentinel node procedure between patients with multifocal and unifocal breast cancer in the EORTC 10981-22023 AMAROS Trial: identification rate and nodal outcome. Eur J Cancer. 2013 Jun;49(9):2093-100. doi: 10.1016/j.ejca.2013.02.017. Epub 2013 Mar 19. PMID 23522754